CLINICAL TRIAL: NCT03701737
Title: Study of Eating Behaviour and Sense of Taste Before and After Treatment With Nocturnal Continuous Positive Airway Pressure in Overweight Patients With Obstructive Sleep Apnoea Syndrome.
Brief Title: Study of Eating Behaviour and Sense of Taste Before and After Treatment With Nocturnal Continuous Positive Airway Pressure in Overweight Patients With Obstructive Sleep Apnea Syndrome.
Acronym: GOUSAS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GEORGES APJ 2017
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Obstructive Sleep Apnoea Syndrome
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — * VAS on the feeling of hunger
  * Evaluation of food wanting by the Finlayson test
  * PREFQUEST Questionnaire
  * 24-hour food recall
  * Stunkard Questionnaire
  * Measurement of daytime sleepiness by Epworth score
Device: wrist actimeter — Actimeter delivery: it is worn on the wrist for 7 days, 24 hours a day.
Biological: Blood samples — 2 dry tubes of 7 ml of blood collected at each visit for plasma assays (ghrelin, leptin, FGF 21, amino acids including tryptophan, insulin resistance)

SUMMARY:
Obstructive sleep apnea (OSA) is characterized by a repeated partial or complete obstruction of the airway that results in a intermittent hypoxia and sleep disturbance.

A complex and reciprocal link between obesity and OSA exists. On the one hand, obesity is one of the main risk factors for OSA. On the other hand, OSA seems to promote obesity. The changes in sleep patterns that characterize OSA alter energy metabolism and promote weight gain. In particular, OSA is associated with metabolic disturbances, decreased physical activity and changes in energy expenditure resulting in weight gain. OSA is characterized by resistance to leptin which reduces the feeling of satiety and an increase in ghrelin levels which increases the feeling of hunger.

There may be an increase in food intake, but very few studies have looked at this aspect. Our current knowledge is based on simple patient reports of the amount of food consumed per 24 hours.

First-line treatment of OSA is based on continuous positive airway pressure (CPAP) but this approach is not curative and weight loss is encouraged. CAPP could facilitate weight loss by restoring sleep quality. Paradoxically, recent studies show weight gain proportional to the duration of use of CPP. Randomized controlled trials offering apneic patients a return to physical activity and hygiene-dietary rules have shown an improvement in OSA after weight loss.

A better understanding of the influence of OSA and its treatment on the energy balance through food preferences and olfacto-gustatory sensoriality is an essential prerequisite for personalized nutritional management. In the face of unexpected weight gain under CPP, this type of intervention would be all the more beneficial as OSA and obesity are public health problems representing two independent risk factors for cardiovascular morbidity and mortality with increasing incidence.

We hypothesize that the treatment of OSA with CPAP changes food preferences in favour of fatty and sugary high-calorie foods.

ELIGIBILITY:
Inclusion Criteria:

* Patient with moderate to severe OSA (apnea and hypopnea index > 15/h) for whom a CPAP is indicated
* Obese patient (body mass index > 30 kg/m2)
* Adult Patient
* Patient who has given oral consent
* Patient speaks and reads French
* Patient affiliated to a the national health insurance system

Exclusion Criteria:

* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a measure to judiciary protection
* Pregnant, parturient or breastfeeding woman
* Major unable or unwilling to consent
* Psychiatric, cognitive or neurological disorders making it impossible to assess food preferences
* Eating disorders (anorexia, bulimia)
* Patient suffering from an acute infection, progressive cancer or under treatment interfering with taste (anti-cancer, antibiotics...)
* Patient consuming alcohol daily
* Patient who smokes actively or has quit for less than 6 months
* Weight change of more than 10% in body weight in the six months before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting a physician
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
food wanting by Finlayson's standardized computerized test | Day 0 and 45

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France